CLINICAL TRIAL: NCT04427865
Title: Efficacy of Lactoferrin as a Preventive Agent for Healthcare Workers Exposed to COVID-19
Brief Title: Utility of Lactoferrin as a Preventive Agent for Healthcare Workers Exposed to COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal Esmat, Professor of Endemic Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CUKA-002
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin prophylaxis (Experimental): 200 mg oral lactoferrin daily
  Interventions: Drug: prophylactic lactoferrin daily
- Control group (No Intervention)

INTERVENTIONS:
Drug: prophylactic lactoferrin daily — 200 mg oral lactoferrin daily
  Arms: Lactoferrin prophylaxis

SUMMARY:
COVID 19, which probably started from zoonotic transmission related to crowded markets in China was announced as a pandemic by the WHO on 11 March 2020.

There is currently no clinically proven specific antiviral agents available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

Since its discovery, lactoferrin and its related peptides are considered non-specific host defense molecules against a broad range of viruses including SARS-CoV, which is closely related to SARS-CoV-2 that causes COVID-19. Besides reducing viral entry, lactoferrin can also suppress virus replication after the viral entry and has an immunomodulatory effect that can prevent the cytokine storm associated with COVID-19.

The aim of our study is to assess the safety and efficacy of lactoferrin within the context of SARS-CoV-2 and propose the possibility of supplemental lactoferrin as a potential preventive drug for healthcare workers exposed to SARS-CoV-2.

DETAILED DESCRIPTION:
In December, 2019, an outbreak of pneumonia with unknown cause occurred in Wuhan city, in China. On January 7th, the scientists succeeded to isolate a novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). WHO nominated it as coronavirus disease 2019 (COVID-19) in February, 2020. COVID-19 has a wide clinical spectrum ranging between asymptomatic infection, mild upper respiratory tract symptoms, and severe viral pneumonia that may result in respiratory failure and finally death. There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

Lactoferrin is a highly conserved pleiotropic iron-binding 80-kDa glycoprotein of the transferrin family that is expressed and secreted by glandular cells and found in most body fluids with especially high concentrations in mammalian milk. Since its discovery, lactoferrin and its related peptides are mainly considered to be important non-specific host defense molecules against a broad range of viruses including SARS-CoV, which is closely related to SARS-CoV-2 that causes COVID-19. Lactoferrin has been found to experimentally inhibit viral entry in murine coronavirus, and human coronaviruses hCOV-NL63 and pseudotyped SARS-CoV. Given the homology of SARS-CoV and SARS-CoV-2 spike protein structures, as well as both viruses depending on the same ACE2 receptor for cell entry, it is likely that lactoferrin can inhibit SARS-CoV-2 invasion as in the case of SARS-CoV. Besides reducing viral entry, lactoferrin can also suppress virus replication after the viral entry as in the case of HIV.

Another major aspect of lactoferrin bioactivity relates to its immunomodulatory and anti-inflammatory functions. Current thinking suggests that mortality from COVID-19 is not simply due to viral infection but is a result of a cytokine storm associated with hyper-inflammation leading to acute respiratory distress and subsequent mortality. A cytokine profile in severe COVID-19 cases is characterized by increases in cytokines and acute phase reactants such as interleukin IL-6, tumor necrosis factor-a (TNFa) and ferritin. In this regard, lactoferrin was demonstrated to reduce IL-6, TNF a, and downregulate ferritin in experimental settings simulating sepsis.

In this study, we aim to study the antiviral properties and immunomodulatory mechanisms of lactoferrin within the context of its potential applications against SARS-CoV-2 and propose the possibility of supplemental lactoferrin as a potential preventive agent for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* health care workers at risk of SARS-CoV-2 transmission with no previous diagnosis of SARS-CoV-2 infection
* No symptoms compatible with SARS-CoV-2 (COVID-19) until the date of enrolment in the study.

Exclusion Criteria:

* Known allergy or hypersensitivity to the used medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 | 28 days
  Number of confirmed infections of SARS-CoV-2 in healthcare workers

SECONDARY OUTCOMES:
Severity of disease in confirmed infected participants | 28 days